CLINICAL TRIAL: NCT05329220
Title: Evaluation of the Immunogenicity, Safety, and Tolerability of a Single Dose of ABNCoV2 Vaccine in Adult Subjects Previously Vaccinated for SARS-CoV-2: a Phase 3 Trial in Two Parts
Brief Title: ABNCoV2 Vaccine in Adult Subjects Previously Vaccinated for SARS-CoV-2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bavarian Nordic (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ABNCoV2-03
Record Dates: First submitted 2022-03-25; First posted 2022-04-14 (Actual); Results first posted 2025-02-24 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2024-12

CONDITIONS: COVID-19 Disease
MeSH Terms: interventions — ABNCoV2 vaccine; BNT162 Vaccine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- ABNCoV2 100μg single dose (Experimental): ABNCoV2 100μg single dose
  Interventions: Biological: ABNCoV2
- Comirnaty (Active Comparator): Comirnaty
  Interventions: Biological: Comirnaty

INTERVENTIONS:
Biological: ABNCoV2 — ABNCoV2 100μg single dose
  Arms: ABNCoV2 100μg single dose
Biological: Comirnaty — Comirnaty
  Arms: Comirnaty

SUMMARY:
This trial is composed of a randomized, double-blind, active controlled component (Part A) and an open-label, single-arm component (Part B) conducted in parallel.

Part A is designed to compare vaccination with a single 100 µg dose of ABNCoV2 to a single 30 µg adult booster dose of Comirnaty (active control) in adult subjects who either previously completed primary vaccination (Cohort 1) or have already received 1 booster dose (Cohort 2) of SARS-CoV-2 locally authorized vaccine(s), and whose last locally authorized SARS-CoV-2 vaccination was at least 3 months prior to the screening visit. Subjects will be randomized in a 1:1 ratio to receive either ABNCoV2 or Comirnaty.

Part B is designed to collect ABNCoV2 safety and tolerability data from a larger population of adult subjects, as well as additional immunogenicity data from a subset. Part B involves vaccination with the same single 100 µg dose of ABNCoV2 in the same population of adult subjects as the randomized component, and subjects will similarly be enrolled into 2 cohorts according to whether they have completed primary vaccination only or primary plus booster vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years at screening.
* Documented, previous completion of a primary vaccination regimen with locally authorized SARS-CoV-2 vaccine(s) or completion of primary plus 1 boost vaccination, with last vaccination at least 3 months before screening. "Locally authorized" SARS-CoV-2 vaccines are those that have received market approval or emergency use authorization in the country of enrollment.
* Absence of acute medical illness, significant physical exam findings, or laboratory abnormalities, as determined by the investigator.
* Informed consent, provided by the subject prior to performance of any trial-specific procedures; the subject has read, signed, and dated an informed consent form (ICF), having been advised of the risks and benefits of the trial in a language understood by the subject.
* Body mass index (BMI) ≥18.5 and <40.
* For female subjects of childbearing potential (WOCBP) and male subjects who are sexually active with a WOCBP, agreement to use an effective method of birth control from at least 30 days prior to administration of the vaccine until 30 days after the vaccination. A woman is considered of childbearing potential unless post-menopausal (defined as ≥12 months without a menstrual period at screening) or surgically sterilized (bilateral oophorectomy, bilateral tubal ligation, hysterectomy). Acceptable contraception methods are restricted to abstinence (only acceptable if refraining from heterosexual intercourse during the period of 30 days prior to administration of the vaccine until 30 days after the vaccination), double barrier contraceptives, vasectomy, intrauterine contraceptive devices, or licensed hormonal products.
* For WOCBP, a negative serum pregnancy test at screening.
* Negative tests for human immunodeficiency virus antibody (anti HIV), hepatitis B surface antigen (HBsAG), and antibody to hepatitis C virus (HCV).

Exclusion Criteria:

* History of COVID 19 infection within the last 3 months before screening.
* Previous vaccination with a SARS-CoV-2 vaccine other than those mentioned in inclusion criterion #2.
* Positive test for SARS-CoV-2 infection at screening.
* Breastfeeding with intent to continue.
* Acute or chronic medical condition that, in the opinion of the investigator, would render the trial procedures unsafe or would interfere with the evaluation of the responses.
* History of myocarditis or pericarditis.
* History of or active autoimmune disease. History of Guillain-Barré syndrome or Reye's syndrome. Persons with vitiligo or thyroid disease taking thyroid replacement are not excluded.
* Known or suspected impairment of immunologic functions including, but not limited to, known immunodeficiency syndrome.
* History of malignancy other than squamous cell or basal cell skin cancer, unless there has been surgical excision at least 6 months prior to screening that is considered to have achieved cure. Subjects with history of skin cancer must not be vaccinated at the previous tumor site.
* Laboratory parameters (such as complete blood count, serum biochemistry including aspartate aminotransferase [AST], alanine amino transferase [ALT], alkaline phosphokinase [ALP], bilirubin, or creatinine values), pulse rate, or blood pressure outside normal range at screening and deemed clinically relevant by the investigator.
* Clinically significant mental disorder not adequately controlled by medical treatment.
* Active or recent history (within 6 months before screening) of chronic alcohol abuse, or illicit drug abuse.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine.
* History of anaphylaxis or severe allergic reaction to any vaccine.
* History of any vaccinations or plan to receive any vaccinations with a live vaccine within 30 days prior to or after trial vaccination.
* History of any vaccinations or plan to receive any vaccinations with a non-live vaccine within 14 days prior to or after trial vaccination.
* Recent blood donation (including platelets, plasma and red blood cells) within 4 weeks prior to screening, or planned blood donations during the active phase of the trial.
* Chronic systemic administration (defined as more than 14 days) of >5 mg prednisone (or equivalent)/day, or any other immune-modifying drugs during a period starting 3 months prior to administration of the vaccine and ending 4 weeks after vaccination. The use of topical, inhaled, ophthalmic and nasal glucocorticoids is allowed.
* History of organ transplantation, whether or not accompanied by chronic immunosuppressive therapy.
* Administration or planned administration of immunoglobulins and/or any blood products during a period starting 3 months prior to administration of the vaccine and ending 4 weeks after vaccination. Receipt of packed red blood cells given for an emergency indication in an otherwise healthy person, and not required as ongoing treatment is not exclusionary (for example packed red blood cells given in emergency during an elective surgery).
* Use of any investigational or non-registered drug or vaccine other than the trial vaccine within 30 days preceding the administration of trial vaccine, or planned administration of such a drug or vaccine throughout the trial.
* Involvement in this trial as site personnel.
* Known bleeding disorder that, in the opinion of the investigator, would contraindicate intramuscular injection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4205 (Actual)
Dates: Start 2022-08-30 (Actual); Primary Completion 2023-03-15 (Actual); Study Completion 2023-10-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leo James, MD, Study Director — Bavarian Nordic
Locations (57):
- United States (44):
  - Achieve Clinical Research LLC d/b/a Accel Research Sites, Birmingham, Alabama
  - Arizona Clinical Trials, Mesa, Arizona
  - Tucson Neuroscience Research - M3 WR, Tucson, Arizona
  - Wr-Pri, Llc, Los Alamitos, California
  - PRI, LLC - Newport Beach - M3 WR, Newport Beach, California
  - FOMAT Medical Research, Oxnard, California
  - Women's Healthcare Research Corporation, San Diego, California
  - Medical Center For Clinical Research, San Diego, California
  - Tekton Research, Fort Collins, Colorado
  - Clinical Site Partners, Leesburg, Florida
  - Accel Research Sites, Maitland, Florida
  - Suncoast Research Group LLC, Miami, Florida
  - Suncoast Research Associates LLC, Miami, Florida
  - Clinical Site Partners, Miami, Florida
  - TrueBlue Clinical Research, Tampa, Florida
  - Clinical Site Partners, Winter Park, Florida
  - Atlanta Center for Medical Research - CenExel ACMR, Atlanta, Georgia
  - Tekton Research, Chamblee, Georgia
  - Columbus Regional Research Institute at Talbotton, Columbus, Georgia
  - Accel Research Site - NeuroStudies.net, LLC, Decatur, Georgia
  - Mount Vernon Clinical Research, LLC, Sandy Springs, Georgia
  - Meridian Clinical Research, LLC, Savannah, Georgia
  - AES - DRS - Synexus Clinical Research US, Inc., Evansville, Indiana
  - Meridian Clinical Research, Sioux City, Iowa
  - CBH Health - CenExel CBH, Gaithersburg, Maryland
  - Sundance Clinical Research, St Louis, Missouri
  - Meridian Clinical Research , LLC, Grand Island, Nebraska
  - Meridian Clinical Research LLC, Lincoln, Nebraska
  - Quality Clinical Research, Inc., Omaha, Nebraska
  - Meridian Clinical Research, Omaha, Nebraska
  - Meridian Clinical Research, Binghamton, New York
  - Emerging Medical Research, LLC, Durham, North Carolina
  - Carolina Institute for Clinical Research, Fayetteville, North Carolina
  - M3 Wake Research, Inc, Raleigh, North Carolina
  - Meridian Clinical Research, LLC, Cincinnati, Ohio
  - Tekton Research, Edmond, Oklahoma
  - ClinSearch, LLC, Chattanooga, Tennessee
  - Tekton Research, Austin, Texas
  - Tekton Research, Beaumont, Texas
  - Global Medical Research, Dallas, Texas
  - Ventavia Research Group, Fort Worth, Texas
  - Ventavia Research Group, Houston, Texas
  - DM Clinical Research, Sugar Land, Texas
  - Meridian Clinical Research - Family Practice, Portsmouth, Virginia
- Belgium (5):
  - Instituut voor Tropische Geneeskunde, Antwerp
  - Centrum voor de evaluatie van vaccinaties, Edegem
  - Private Practice Dr Jean Benoit Martinot, Erpent
  - Centrum voor vaccinologie (CEVAC), Ghent
  - Office of Marc De Meulemeester, Gozée
- Denmark (8):
  - Aalborg Universitetshospital, Aalborg
  - Aarhus Universitetshospital, Aarhus
  - Bispebjerg Hospital, Afdeling for Lunge- og Infektionssygdomme, Copenhagen
  - Regionshospitalet Gødstrup, Medicinsk afdeling, Klinik for Infektionssygdomme, Herning
  - Nordsjællands Hospital, Hillerød, Lunge- og Infektionsmedicinsk Afdeling, Hillerød
  - Hvidovre Hospital, Infektionsmedicinsk afd., Hvidovre
  - Odense Universitetshospital, Q, Infektionsmedicinsk Afdeling, Odense
  - Sjællands Universitetshospital, Roskilde

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: At least 500 subjects were to be enrolled into Part A of this trial, and approximately 3000 subjects were to be enrolled into Part B. Enrollment for Part A and Part B occurred simultaneously and enrollment was based on prior SARS-CoV-2 experience, with Cohort 1 including an authorized primary vaccination regimen; and Cohort 2 including an authorized primary vaccination regimen with a booster vaccination.
Pre-assignment Details: Three subjects were randomized but were withdrawn prior to receiving study product. One subject withdrew consent and two subjects were randomized in error and withdrawn due to not meeting inclusion/exclusion criteria.
Groups:
- Part A Cohort 1 ABNCoV2; Part B Cohort 1 ABNCoV2: Subjects who previously completed primary vaccination 100ug ABNCoV2 by subcutaneous injection on Day 1
- Part A Cohort 1 Comirnaty: Subjects who previously completed primary vaccination 30ug Comirnaty by subcutaneous injection on Day 1
- Part A Cohort 2 ABNCoV2; Part B Cohort 2 ABNCoV2: Subjects who previously completed primary vaccination plus 1 booster 100ug ABNCoV2 by subcutaneous injection on Day 1
- Part A Cohort 2 Comirnaty: Subjects who previously completed primary vaccination plus 1 booster 30ug Comirnaty by subcutaneous injection on Day 1
Period: Active Trial Period
Arm/Group | Part A Cohort 1 ABNCoV2 | Part A Cohort 1 Comirnaty | Part A Cohort 2 ABNCoV2 | Part A Cohort 2 Comirnaty | Part B Cohort 1 ABNCoV2 | Part B Cohort 2 ABNCoV2
Started | 34 | 34 | 277 | 277 | 1438 | 2145
Completed | 34 | 34 | 277 | 276 | 1390 | 2098
Not Completed | 0 | 0 | 0 | 1 | 48 | 47
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 32 | 28
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 2 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 1 | 3
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 12 | 13
Not completed — SPONSOR GUIDANCE DUE TO SUBJECT'S CHANGE IN SCHEDULE WITH TRAVELING OUT OF THE COUNTRY | 0 | 0 | 0 | 0 | 0 | 1
Not completed — THE PARTICIPANT HAD TO BE DROPPED FROM THE STUDY AS THEY WERE UNABLE TO CONTINUE. | 0 | 0 | 0 | 0 | 0 | 1
Not completed — SUBJECT WAS OOW | 0 | 0 | 0 | 0 | 0 | 1
Period: Follow-up Period
Arm/Group | Part A Cohort 1 ABNCoV2 | Part A Cohort 1 Comirnaty | Part A Cohort 2 ABNCoV2 | Part A Cohort 2 Comirnaty | Part B Cohort 1 ABNCoV2 | Part B Cohort 2 ABNCoV2
Started (Subject could participate in follow-up even if not completing the active trial period.) | 34 | 34 | 277 | 277 | 1438 | 2144
Completed | 34 | 33 | 272 | 273 | 1285 | 2009
Not Completed | 0 | 1 | 5 | 4 | 153 | 135
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 2 | 1
Not completed — Death | 0 | 0 | 1 | 1 | 0 | 1
Not completed — Lost to Follow-up | 0 | 1 | 2 | 2 | 113 | 89
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 2 | 2
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 1 | 34 | 35
Not completed — PATIENT WORKS IN AUSTRALIA SINCE JUNE2023 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — SUBJECT WAS GOING OUT OF TOWN FOR AN EXTENDED PERIOD OF TIME | 0 | 0 | 0 | 0 | 1 | 0
Not completed — SUBJECT NON-COMPLIANCE | 0 | 0 | 0 | 0 | 1 | 0
Not completed — SUBJECT MOVED OUT OF TOWN | 0 | 0 | 0 | 0 | 0 | 1
Not completed — EARLY TERMINATION | 0 | 0 | 0 | 0 | 0 | 1
Not completed — SUBJECT HAD BUT DID NOT COMPLETE THEIR FINAL VISIT WITHIN 14 DAYS BEFORE THE V1 + 182 DAYS | 0 | 0 | 0 | 0 | 0 | 2
Not completed — DROPPED | 0 | 0 | 0 | 0 | 0 | 1
Not completed — DROPPED DUE TO BEING UNABLE TO CONTINUE IN THE TRIAL. | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: "All subjects who received at least one vaccination with ABNCoV2 at any time during the trial. "
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A Cohort 1 ABNCoV2 | Part A Cohort 1 Comirnaty | Part A Cohort 2 ABNCoV2 | Part A Cohort 2 Comirnaty | Part B Cohort 1 ABNCoV2 | Part B Cohort 2 ABNCoV2 | Total
Number analyzed (Participants) | 34 | 34 | 277 | 277 | 1438 | 2145 | 4205
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 34 | 34 | 247 | 249 | 1147 | 1356 | 3067
  >=65 years | 0 | 0 | 30 | 28 | 291 | 789 | 1138
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.4 (13.44) | 32.2 (11.67) | 42.8 (16.4) | 41.8 (15.91) | 48.2 (15.6) | 54.5 (15.73) | 50.4 (16.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 12 | 133 | 135 | 813 | 1210 | 2318
  Male | 19 | 22 | 144 | 142 | 625 | 935 | 1887
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 00 | 1 | 2 | 3 | 623 | 593 | 1222
  Not Hispanic or Latino | 34 | 33 | 274 | 274 | 795 | 1523 | 2933
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 20 | 29 | 50
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 6 | 17 | 23
  Asian | 0 | 0 | 2 | 1 | 27 | 59 | 89
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 3 | 3
  Black or African American | 0 | 0 | 0 | 1 | 439 | 469 | 909
  White | 33 | 34 | 272 | 273 | 911 | 1521 | 3044
  More than one race | 0 | 0 | 0 | 1 | 14 | 28 | 43
  Unknown or Not Reported | 1 | 0 | 3 | 1 | 41 | 48 | 94
Region of Enrollment [Number; unit: participants]
  Belgium | 24 | 26 | 161 | 167 | 0 | 0 | 378
  United States | 0 | 0 | 0 | 0 | 1438 | 2145 | 3583
  Denmark | 10 | 8 | 116 | 110 | 0 | 0 | 244

OUTCOME MEASURES:

1. Primary Outcome: Neutralizing Antibody Titers Against the SARS-CoV-2 Index Virus (Wuhan Wild Type Isolate) at 2 Weeks After Trial Vaccination
Description: The primary endpoint was SARS-CoV-2 index virus (Wuhan wild type isolate) neutralizing antibodies assessed at 2 weeks after trial vaccination, for subjects in the Immunogenicity Analysis Sets in Part A Cohort 1 (adult subjects who previously completed primary vaccination at least 3 months prior to the screening visit) and Part A Cohort 2 (adult subjects who have completed primary vaccination and have received 1 booster vaccination).
Time Frame: 2 weeks after the single trial vaccination occurring on Day 1
Population: All subjects who are in the Safety Analysis Set, have at least a baseline and 1 post-vaccination neutralizing antibody result, and have neither intercurrent events indicative of SARSCoV2 infection nor received a booster for SARSCoV2 outside of the trial within 2 weeks of vaccination. Subjects with protocol deviations substantially affecting the immunogenicity outcomes were excluded from this analysis set.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Part A Cohort 1 ABNCoV2 | Part A Cohort 1 Comirnaty | Part A Cohort 2 ABNCoV2 | Part A Cohort 2 Comirnaty
Number analyzed (Participants) | 34 | 33 | 267 | 261
titer | 1018.1 [621.1 to 1669.0] | 1060.6 [708.2 to 1588.3] | 1259.0 [1125.3 to 1408.4] | 1619.6 [1485.9 to 1765.4]
Statistical Analysis 1: Comparison: Part A Cohort 1 ABNCoV2 vs Part A Cohort 1 Comirnaty; Formal hypothesis testing was performed due to having at least 400 evaluable subjects with primary endpoint data available at baseline and at 2 weeks after trial vaccination. The null hypothesis is that ABNCoV2 is inferior to Comirnaty and will be rejected if the ratio of the GMTs for ABNCoV2 versus Comirnaty is within the non-inferiority margin of 0.67; that is, the lower bound of the 2-sided 97.5% CI of the GMT ratio is >=0.67; Test type: Non-Inferiority — The success criterion for the null hypothesis that ABNCoV2 is inferior to Comirnaty will be rejected if the ratio of the GMTs for ABNCoV2 versus Comirnaty is within the non-inferiority margin of 0.67; that is, the lower bound of the 2-sided 97.5% CI of the GMT ratio is >=0.67; p = 0.6350, Mixed Models Analysis — P-value corresponds to Cohort 1 ABNCoV2 comparison to Cohort 1 Comirnaty; A generalized linear model with age and baseline results included as covariates was used to compare between the vaccination groups; Geometric Mean Ratio = 0.89, 97.5% CI 2-sided [0.50 to 1.57]
Statistical Analysis 2: Comparison: Part A Cohort 2 ABNCoV2 vs Part A Cohort 2 Comirnaty; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.0002, Mixed Models Analysis — P-value corresponds to Cohort 2 ABNCoV2 comparison to Cohort 2 Comirnaty; [statistical method as in outcome 1, analysis 1]; Geometric Mean Ratio = 0.80, 97.5% CI 2-sided [0.70 to 0.92]

2. Secondary Outcome: Neutralizing Antibody Titers Against the SARS-CoV-2 Variants of Concern (Omicron Variants BA.4/BA.5 and XBB.1.5) at 2 Weeks After Trial Vaccination
Description: The secondary endpoint was SARS-CoV-2 variants of concern (Omicron Variant BA.4/BA.5 and XBB.1.5) pseudovirus or virus neutralizing antibodies assessed at 2 weeks after trial vaccination, for subjects in the Immunogenicity Analysis Sets in Part A Cohort 1 (adult subjects who previously completed primary vaccination at least 3 months prior to the screening visit) and Part A Cohort 2 (adult subjects who have completed primary vaccination and have received 1 booster vaccination.
Time Frame: 2 weeks after the single trial vaccination occurring on Day 1
Population: All subjects who are in the Safety Analysis Set, have at least a baseline and 1 post-vaccination neutralizing antibody result, and have neither intercurrent events indicative of SARSCoV2 infection nor received a booster for SARSCoV2 outside of the trial within 2 weeks of vaccination. Subjects with protocol deviations substantially affecting the immunogenicity outcomes were excluded. Part A Cohort 2 is the only group that met the primary endpoint criteria and are the only results analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Part A Cohort 2 ABNCoV2 | Part A Cohort 2 Comirnaty
Number analyzed (Participants) | 265 | 260
titer
  Omicron Variant BA.4/BA.5 | 17112.6 [14775.8 to 19818.9] | 23506.3 [20794.5 to 26571.7]
  Omicron Variant XBB.1.5 | 54.7 [48.9 to 61.3] | 81.3 [73.1 to 90.4]
Statistical Analysis 1: Comparison: Part A Cohort 2 ABNCoV2 vs Part A Cohort 2 Comirnaty; Formal hypothesis testing was performed due to meeting the primary endpoint success criterion in Cohort 2. The null hypothesis is that ABNCoV2 is inferior to Comirnaty and will be rejected if the ratio of the GMTs for ABNCoV2 versus Comirnaty is within the non-inferiority margin of 0.67; that is, the lower bound of the 2-sided 97.5% CI of the GMT ratio is >=0.67; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.0008, Mixed Models Analysis — P-value corresponds to Cohort 2 ABNCoV2 comparison to Cohort 2 Comirnaty for Omicron variant BA.4/BA.5; [statistical method as in outcome 1, analysis 1]; Geometric Mean Ratio = 0.76, 97.5% CI 2-sided [0.64 to 0.91]
Statistical Analysis 2: Comparison: Part A Cohort 2 ABNCoV2 vs Part A Cohort 2 Comirnaty; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p < 0.0001, Mixed Models Analysis — P-value corresponds to Cohort 2 ABNCoV2 comparison to Cohort 2 Comirnaty for Omicron Variant XBB.1.5; [statistical method as in outcome 1, analysis 1]; Geometric Mean Ratio = 0.69, 97.5% CI 2-sided [0.59 to 0.81]

3. Secondary Outcome: Neutralizing Antibody Titers Against the SARS-CoV-2 Index Virus (Wuhan Wild Type Isolate) at 2 Weeks After Trial Vaccination [Time Frame: 2 Weeks After the Single Trial Vaccination Occurring on Day 1]
Description: The secondary endpoint was SARS-CoV-2 index virus (Wuhan wild type isolate) neutralizing antibodies assessed at 2 weeks after trial vaccination, for subjects in the Immunogenicity Analysis Sets in Part B Cohort 1 (adult subjects who previously completed primary vaccination at least 3 months prior to the screening visit) and Part B Cohort 2 (adult subjects who have completed primary vaccination and have received 1 booster vaccination).
Time Frame: 2 weeks after the single trial vaccination occurring on Day 1
Population: This secondary endpoint was defined in the protocol and originally intended to be performed on the Part B Cohorts. However, based on the assessment of Part A lower neutralizing antibody results versus the comparator it was decided not to analyze the Part B open-label samples. Due to there being no assays performed, there are no assay results to report.
Arm/Group | Part B Cohort 1 ABNCoV2 | Part B Cohort 2 ABNCoV2
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Safety and Tolerability of the ABNCoV2 Vaccine as Measured by the Frequency of Solicited and Unsolicited Adverse Events Occurring During or After the Trial Vaccination.
Description: The number and percent of subjects who report:
  * SAEs or AESIs assessed as related to trial vaccine during the entire trial period, which includes both the active trial phase and follow-up.
  * Grade 3 or higher AEs assessed as related to trial vaccine in the 8 day period starting with the day of vaccination.
  * SAEs, AESIs or MAAEs, regardless of relationship, during the active trial phase.
  * SAE, AESI or MAAEs, regardless of relationship, during the entire trial period.
  * Grade 3 or higher AEs assessed as related to trial vaccine during the active trial phase.
  * Solicited local AEs in the 8 day period starting with the day of vaccination.
  * Solicited general AEs in the 8 day period starting with the day of vaccination.
  Solicited event grading based on FDA 2007 Guidance for industry: toxicity grading scale for healthy adult and adolescent volunteers enrolled in preventive vaccine clinical trials, where Grade 1 is Mild and Grade 4 is Life-Threatening and the worst outcome.
Time Frame: Active trial period is from vaccination until 28 to 35 days after vaccination. Entire trial period is from vaccination until 182 to 196 days after vaccination. Solicited events are reported if occurring within 8 days following vaccination.
Population: All subjects who received at least one vaccination with ABNCoV2 at any time during the trial.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A Cohort 1 ABNCoV2 | Part A Cohort 1 Comirnaty | Part A Cohort 2 ABNCoV2 | Part A Cohort 2 Comirnaty | Part B Cohort 1 ABNCoV2 | Part B Cohort 2 ABNCoV2
Number analyzed (Participants) | 34 | 34 | 277 | 277 | 1438 | 2145
Participants
  Related SAEs during Entire Trial Period | 0 | 0 | 0 | 0 | 0 | 0
  Related AESIs during Entire Trial Period | 0 | 0 | 3 | 0 | 6 | 7
  Related Grade 3 or Higher AEs within 8 Days of Vaccination | 7 | 2 | 28 | 24 | 164 | 188
  SAE, AESI, or MAAE during Active Trial Period | 1 | 3 | 42 | 30 | 96 | 204
  SAE, AESI, or MAAE during Entire Trial Period | 6 | 6 | 85 | 78 | 192 | 442
  Related Grade 3 or Higher AEs during Active Trial Period | 7 | 3 | 35 | 34 | 218 | 272
  Solicited Local AE within 8 Days of Vaccination | 28 | 30 | 238 | 236 | 810 | 1269
  Solicited Systemic AE within 8 Days of Vaccination | 23 | 17 | 185 | 170 | 715 | 1139

ADVERSE EVENTS:
Time Frame: Overall trial from vaccination through final follow-up visit occurring between Day 182 and Day 196 after vaccination.
Arm/Group | Part A Cohort 1 ABNCoV2 | Part A Cohort 1 Comirnaty | Part A Cohort 2 ABNCoV2 | Part A Cohort 2 Comirnaty | Part B Cohort 1 ABNCoV2 | Part B Cohort 2 ABNCoV2
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/34 | 1/277 | 1/277 | 0/1438 | 1/2145
Serious Adverse Events (participants affected / at risk) | 2/34 | 0/34 | 3/277 | 7/277 | 23/1438 | 49/2145
Other Adverse Events (participants affected / at risk) | 6/34 | 4/34 | 40/277 | 47/277 | 36/1438 | 125/2145
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A Cohort 1 ABNCoV2 (N=34) | Part A Cohort 1 Comirnaty (N=34) | Part A Cohort 2 ABNCoV2 (N=277) | Part A Cohort 2 Comirnaty (N=277) | Part B Cohort 1 ABNCoV2 (N=1438) | Part B Cohort 2 ABNCoV2 (N=2145)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Abdominal wall abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthritis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Helicobacter infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Large intestine infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Liver abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pelvic inflammatory disease (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Perirectal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dengue fever (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intervertebral discitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cerebral infarction (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myocarditis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Spinal cord injury cervical (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wound necrosis (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Acoustic neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Brain cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Small cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 3 (3)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
End stage renal disease (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Obstructive nephropathy (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bipolar disease (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Delirium tremens (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Major depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Completed suicide (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peptic ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arterial occlusive disease (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood loss anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Abnormal uterine bleeding (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pelvic organ prolapse (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vertigo positional (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Systemic inflammatory response syndrome (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Astrovirus test positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A Cohort 1 ABNCoV2 (N=34) | Part A Cohort 1 Comirnaty (N=34) | Part A Cohort 2 ABNCoV2 (N=277) | Part A Cohort 2 Comirnaty (N=277) | Part B Cohort 1 ABNCoV2 (N=1438) | Part B Cohort 2 ABNCoV2 (N=2145)
COVID-19 (Infections and infestations) | 1 (1) | 1 (1) | 17 (17) | 14 (14) | 36 (36) | 125 (125)
Nasopharyngitis (Infections and infestations) | 2 (2) | 0 (0) | 15 (15) | 21 (21) | 5 (5) | 13 (13)
Pharyngitis (Infections and infestations) | 1 (1) | 2 (2) | 2 (2) | 3 (3) | 3 (3) | 5 (5)
Headache (Nervous system disorders) | 3 (3) | 1 (1) | 11 (11) | 10 (11) | 11 (11) | 16 (17)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution/Investigator agree to submit any proposed publication or presentation to Sponsor for review at least 60 days prior to submitting any such proposed publication to a publisher or proceeding with such proposed presentation. Sponsor shall have the right to require Institution/Investigator to remove specifically identified Confidential Information and/or to delay the proposed publication or presentation for an additional 60 days to enable Sponsor to seek patent protection for Inventions.

DOCUMENTS (2):
  • Study Protocol (2023-06-30): https://cdn.clinicaltrials.gov/large-docs/20/NCT05329220/Prot_000.pdf
  • Statistical Analysis Plan (2023-05-24): https://cdn.clinicaltrials.gov/large-docs/20/NCT05329220/SAP_001.pdf